CLINICAL TRIAL: NCT06770283
Title: Research on the Prevention and Treatment of Liver Fibrosis/Cirrhosis with Spirulina Tablets and Its Mechanisms
Brief Title: Spirulina Tablets Treat Liver Fibrosis/Cirrhosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-1239
Record Dates: First submitted 2024-12-29; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Liver Cirrhosis
Keywords: Liver cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- placebo (Placebo Comparator): The control group will receive an equivalent dose of maltodextrin for at least 3 weeks.
  Interventions: Dietary Supplement: Maltodextrin (Placebo)
- Spirulina treatment (Active Comparator): In the Spirulina tablet intervention group, patients will receive oral Spirulina tablet treatment (2g/day) for at least 3 weeks before liver transplantation.
  Interventions: Dietary Supplement: Spirulina tablet

INTERVENTIONS:
Dietary Supplement: Spirulina tablet — In the Spirulina tablet intervention group, patients will receive oral Spirulina tablet treatment (2g/day) for at least 3 weeks before liver transplantation.
  Arms: Spirulina treatment
Dietary Supplement: Maltodextrin (Placebo) — In the control group, patients will receive oral maltodextrin tablet treatment (2g/day) for at least 3 weeks before liver transplantation.
  Arms: placebo

SUMMARY:
Spirulina (Spirulina platensis, SP) is a nutrient-rich blue-green algae that has been widely studied and applied in various health fields. Its main components include spirulina polysaccharide proteins, amino acids, vitamins, and minerals, especially the eight essential amino acids that the human body cannot synthesize on its own. Spirulina is also rich in minerals such as iron, calcium, and zinc, which makes it beneficial in the prevention and treatment of several diseases. Research has shown that spirulina has potential therapeutic effects in combating tumors, obesity, diabetes, cardiovascular diseases, and anemia. In 2020, the National Health Commission of the People's Republic of China classified it as a health food supplement.

Hepatic fibrosis (HF) is a process of chronic liver disease caused by excessive repair responses to liver tissue injury due to various factors. As the fibrosis progresses, extracellular matrix in the liver accumulates, forming scar tissue that gradually replaces the normal liver parenchyma. Eventually, these pathological changes can lead to cirrhosis, portal hypertension, and even primary hepatocellular carcinoma (HCC), which may result in liver failure. Therefore, hepatic fibrosis is considered a critical precursor to cirrhosis and liver cancer.

In 2007, Elsharkawy and colleagues proposed the "hepatitis-fibrosis-liver cancer axis" theory, which emphasized that timely treatment of hepatic fibrosis is crucial to controlling the development of cirrhosis and liver cancer. However, modern medicine has yet to discover specific drugs for treating hepatic fibrosis or cirrhosis. The etiology of hepatic fibrosis is complex, involving various cellular and molecular mechanisms, thus making the in-depth study of its pathogenesis and the development of new treatments particularly urgent.

As the understanding of hepatic fibrosis continues to deepen, increasing attention is being given to the potential of natural products or health supplements in preventing and treating hepatic fibrosis. Spirulina, as a natural product with multiple biological activities, may become a promising direction for exploring new treatments for hepatic fibrosis due to its immune-regulating, antioxidant, and anti-inflammatory effects. Through further clinical and experimental research, spirulina may offer a new complementary treatment option for hepatic fibrosis.

ELIGIBILITY:
Inclusion Criteria for Patients:

* Diagnosed with liver fibrosis or cirrhosis.
* Patients scheduled for liver transplantation with a waiting time of more than 3 weeks.
* Adults aged 18 to 75 years.
* Willing to participate in the study and sign an informed consent form.
* No acute diseases or significant exacerbation of symptoms in the 4 weeks prior to enrollment.

Exclusion Criteria:

* Patients with severe comorbidities.
* Patients allergic to Spirulina tablets.
* Patients with a history of severe mental illness that could affect treatment adherence.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-12-26 (Actual); Primary Completion 2026-12-26 (Estimated); Study Completion 2026-12-26 (Estimated)

PRIMARY OUTCOMES:
single-cell and/or transcriptome sequencing | through study completion, an average of 1 year
  Prospective collection of patient fecal samples will be performed with the following sampling frequency: one sample will be collected on Day 0 before treatment, and another sample will be collected after the treatment is completed. These samples will undergo metagenomic sequencing of the gut microbiome. Prospective collection of liver tissue samples from liver transplant surgeries of patients with liver fibrosis/cirrhosis will be done, with each sample approximately 1 cm³ in size. The samples will be immediately stored at -80°C for single-cell and/or transcriptome sequencing.

SECONDARY OUTCOMES:
Evaluation of intestinal flora | through study completion, an average of 1 year
  Prospective collection of patient fecal samples will be performed with the following sampling frequency: one sample will be collected on Day 0 before treatment, and another sample will be collected after the treatment is completed. These samples will undergo metagenomic sequencing of the gut microbiome.
  High-throughput sequencing is used to sequence the 16S rDNA of prokaryotes, with the aim of detecting the microbial composition and abundance in the samples.

CONTACTS AND LOCATIONS:
Locations (1):
- 2 nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No